CLINICAL TRIAL: NCT03045965
Title: Hysterectomy and Opportunistic Salpingectomy
Acronym: HOPPSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LUA-HTA-2016:86; VGFOUREG-650491 (Other Grant/Funding Number: Vastra Gotaland Region)
Record Dates: First submitted 2017-01-16; First posted 2017-02-08 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer; Complication
Keywords: Salpingectomy; Hysterectomy; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Salpingectomy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking of the intervention is planned to include the one-year follow-up of menopausal symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salpingectomy (Experimental): Concomitant salpingectomy at the time of hysterectomy for a benign reason
  Interventions: Procedure: Salpingectomy
- No salpingectomy (No Intervention): No salpingectomy at the time of hysterectomy for a benign reason

INTERVENTIONS:
Procedure: Salpingectomy — The intervention is a routine salpingectomy, performed laparoscopically, through laparotomy or vaginally.
  Arms: Salpingectomy

SUMMARY:
HOPPSA is a register based randomized controlled trial (R-RCT), with the objective to examine if opportunistic salpingectomy compared with no salpingectomy, at the time of hysterectomy for a benign reason

* has no increased risk of complications
* has no negative side effects on ovarian function and subsequent cardiovascular disease or incidence of fractures
* implies reduced risk of subsequent ovarian cancer Randomization and follow-up will be conducted within national registers.

DETAILED DESCRIPTION:
High grade serous ovarian cancer, the most fatal subtype, may originate in the fimbriae of the Fallopian tubes. This theory has led to the idea of opportunistic salpingectomy as a way of decreasing the risk of epithelial ovarian cancer (EOC). HOPPSA is a national register-based RCT, with randomization and follow-up in The Swedish National Quality Register of Gynecological Surgery (Gyn/Op).

HOPPSA aims to study if opportunistic salpingectomy is safe, and if it can reduce the risk of EOC.

PICO P (patients). Women <55 years, undergoing hysterectomy due to a benign reason I (intervention). Bilateral salpingectomy at the time of hysterectomy C (comparison). No salpingectomy O (outcomes). Primary short term: surgical complications reported according to Clavien-Dindo at 8 weeks post-operatively Intermediate term: change in menopausal symptoms from baseline to 1 year, assessed with Menopause Rating Scale Long term: ovarian cancer assessed through the National Cancer Register Recruitment of 4400 patients is estimated to take 4-6 years depending on the participation rate of the Swedish gynecological clinics. Data retrieval from GynOp on short and intermediate term outcomes, requiring smaller sample sizes, will be done at the end of the recruitment period. If these results, ready available when the study recruitment is closed, show that opportunistic salpingectomy does not increase surgical complications and menopausal symptoms, women can be advised to undergo salpingectomy to potentially minimize the future risk of EOC.

ELIGIBILITY:
Inclusion Criteria:

* Planned hysterectomy for a benign reason
* Age < 55 years at randomization
* Willing to be randomized
* Vaginal route may be included if the surgeon is confident with performing vaginal salpingectomy.

Exclusion Criteria:

* Previous bilateral oophorectomy and/or salpingectomy
* Planned oophorectomy and/or salpingectomy (for reasons such as already diagnosed adnexal tumor, known carrier of the breast cancer susceptibility gene (BRCA) 1/2 mutation or Lynch syndrome (hereditary nonpolyposis colorectal cancer))
* Non-understanding of the oral or written study information

Ages: 20 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4400 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2053-12 (Estimated)

PRIMARY OUTCOMES:
Surgical complication - short term primary outcome | Eight weeks post-operative
  Dichotomous outcome, retrieved from any of two sources in the GynOp register: specified question on complications and the Clavien-Dindo classification
Change in menopausal symptom score - intermediate term primary outcome | One year after surgery
  Measured from baseline to one year follow-up, assessed with Menopause Rating Scale (MRS)
Epithelial ovarian cancer - long term primary outcome | 10-30 years after surgery
  The outcome is dichotomous, the diagnosis is classified according to ICD10. Each case with a positive outcome is further described with histopathological types and grade, as well as clinical stage according to International Federation of Gynecology and Obstetrics (FIGO). Assessed through national registers stage according to International Federation of Gynecology and Obstetrics (FIGO). Assessed through national registers

SECONDARY OUTCOMES:
Operative time | At day of surgery
  Continous outcome, registered in minutes
Length of hospital stay | Assessment will be done at discharge from hospital after surgery, including a period up to 8 weeks. a
  Continous outcome, registered in days
Perioperative blood loss | At day of surgery
  Continous outcome, registered in ml
Conversion to other surgical route | At day of surgery
  Dichotomous outcome
Failure rate of salpingectomy at planned vaginal hysterectomy | At day of surgery
  Dichotomous outcome
Prevalence of menopausal symptoms of at least moderate level according to Menopause Rating Scale (MRS) | One and five years after surgery
  Dichotomous outcome based on MRS
Ovarian function, measured as change in anti-Müllerian hormone (AMH) serum level, from baseline | One year after surgery
  Continous outcome, measured in mg/L
Subsequent adnexal surgery, including all surgery engaging salpinges and/or ovaries | At one and up to ten years after surgery
  Dichotomous outcome, accompanied by a description of number and types of surgery performed
Use of Hormone Replacement Therapy (HRT) | At one and up to ten years after surgery
  Dichotomous outcome
Cardiovascular disease | 10-30 years after surgery
  Dichotomous outcome, accompanied by the specific ICD diagnoses
Fractures (primarily radial, vertebral and hip fractures) | 10-30 years after surgery
  Dichotomous outcome, accompanied by the specific ICD diagnoses

CONTACTS AND LOCATIONS:
Overall Officials: Annika Strandell, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Idahl A, Liv P, Darelius A, Collins E, Sundfeldt K, Palsson M, Strandell A. HOPPSA update: changes in the study protocol of Hysterectomy and OPPortunistic SAlpingectomy, a registry-based randomized controlled trial. Trials. 2023 Mar 24;24(1):222. doi: 10.1186/s13063-023-07244-w. PMID 36959664

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03045965/SAP_000.pdf